CLINICAL TRIAL: NCT02840786
Title: Occlusive Disease of Lower Extremity
Brief Title: Clinical Study of Stent Versus Direct Atherectomy to Treat Arteriosclerosis Occlusive Disease of Lower Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuH16
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2016-04

CONDITIONS: Atherosclerosis; Ischemia
Keywords: stents; atherectomy; femoral artery; popliteal artery
MeSH Terms: conditions — Atherosclerosis; Ischemia | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention: Stents (Active Comparator): Stents group
  Interventions: Device: balloon and Stent
- Intervention: Atherectomy (Active Comparator): directional atherectomy group
  Interventions: Device: plaque excision system

INTERVENTIONS:
Device: plaque excision system
  Arms: Intervention: Atherectomy
Device: balloon and Stent
  Arms: Intervention: Stents

SUMMARY:
This is a randomized study comparing stent and plaque excision systems in treatment of Arteriosclerosis occlusive disease of lower extremity (superficial femoral or popliteal artery)

DETAILED DESCRIPTION:
This is a randomized study comparing balloon angioplasty adjunctive stent and plaque excision systems in treatment of Arteriosclerosis occlusive disease of lower extremity (superficial femoral or popliteal artery)

ELIGIBILITY:
Patients were included if they were de novo stenosis>70% or occlusion of the femoropopliteal at least 18 years of age and referred for claudication (Rutherford-Becker class II-III) or critical limb ischemia (Rutherford-Becker class IV-V). They were excluded if they had one or more of the following: 1. Acute or subacute lower limb ischemia; 2. Severe calcification lesions; 3. Total occlusions lesions more significant than 10 cm or total occlusion lesions with a suspicion of subintimal wire recanalization 4. untreated ipsilateral iliac artery stenosis>70%, or the distal runoff artery <1 root; 5. Previously lower extremity intervention or surgical graft artery bypass; 6. Severe renal insufficiency, creatinine level greater than 2.5 mg/dL; 7. The patient's platelet count is less than 100,000/uL, antiplatelet or anticoagulant contraindications to required medications; 8. Patients with immune system diseases or malignant tumours; 9. ongoing active infection 10. decompensated congestive heart failure or acute coronary syndrome; 11. Unwillingness to return for future follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
12-month Primary Patency Rate | 12 months
  systolic velocity ratio >2.4 as measured by Duplex ultrasound.

SECONDARY OUTCOMES:
Technical success | 1 day
  Technical success was defined as residual stenosis less than 30% by final angiography and/or a flow-limiting dissection.
freedom from clinically-driven TLR | 12 months
  it is defined as thefreedom from clinically-driven target lesion revascularization
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization , and significant embolic events, which were defined as causing end-organ damage.
12-month Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided